CLINICAL TRIAL: NCT05390723
Title: Communication in Breast Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Dutch Cancer Society (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, lmvanvliet, Assistant Professor, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N21CPB-IRBd22-103; 2022-01-07-L.M.vanVliet-V1-36 (Other: Dutch Cancer Institute (AVL) and Leiden University)
Record Dates: First submitted 2022-04-12; First posted 2022-05-25 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Communication; Breast Cancer; Quality of Life
Keywords: scripted video-vignette study
MeSH Terms: conditions — Communication; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A single-centre proof-of-principle RCT will be conducted using a scripted video-design. Four different information-videos about chemotherapy's side effects are created in which specific communication is manipulated to assess their effect on patient (psychological/cognitive/physical outcomes. (The investigators cannot yet reveal the manipulation as it would influence our participants)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- video 1 (Experimental): The investigators cannot yet reveal the specific communication that will be manipulate, as this might influence participant outcomes.
  Interventions: Behavioral: Communciation intervention
- video 2 (Experimental): The investigators cannot yet reveal the specific communication that will be manipulate, as this might influence participant outcomes.
  Interventions: Behavioral: Communciation intervention
- video 3 (Experimental): the investigators cannot yet reveal the specific communication that will be manipulate, as this might influence participant outcomes.
  Interventions: Behavioral: Communciation intervention
- video 4 (Experimental): the investigators cannot yet reveal the specific communication that will be manipulate, as this might influence participant outcomes.
  Interventions: Behavioral: Communciation intervention

INTERVENTIONS:
Behavioral: Communciation intervention — The investigators cannot reveal the manipulated communication as this might influence participant outcomes.

SUMMARY:
The investigators will create 4 information-video's about chemotherapy side-effects in curative breast cancer care. The communication is manipulated in the four videos. Participants will watch the video before the first chemotherapy and complete questionnaires before and after viewing the video and after chemotherapy 1,2 and 4. (The investigators cannot yet reveal the manipulation as it would influence the participants)

DETAILED DESCRIPTION:
NA, the investigators cannot yet reveal the manipulation as it would influence the participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) female breast cancer patients
* Chemo-naïve patients
* Scheduled in for curative neo-adjuvant chemotherapy: Four courses of AC chemotherapy (all combinations of AC + other chemotherapy courses are eligible)
* Cognitively able to fill out an online questionnaire
* Having internet access
* Sufficient command of the Dutch language
* pre-chemo no previous treatment or pre-chemo breast-conserving surgery and radiotherapy (WLE patients)

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | Day 0 (day before chemo 1), day 7-10 (week after chemo 1), day 21-23 (week after chemo 2), and day 52-54 (10 days after chemo 4). (This might be subject to change in cases where the days of the chemo therapy are changed
  measuring the change in anxiety measured using a shortened version of the State-Trait Anxiety Inventory (STAI-S)

SECONDARY OUTCOMES:
socio-demographics | Day 0 (day before chemo 1)
  measuring the change in age, SES, education age, SES, education (7 questions)
information needs | Day 0 (day before chemo 1)
  coping infromation needs ( 2 questions)
anxiety | trait: Day 0 (day before chemo 1), current: Day 0 (day before chemo 1), day 7-10 (week after chemo 1), day 21-23 (week after chemo 2), and dday 52-54 (10 days after chemo 4).
  measuring the change in anxiety trait (20 questions) and current anxiety (1 question)
side effects (expected and experienced) | expected: Day 0 (day before chemo 1); experienced: day 7-10 (week after chemo 1), day 21-23 (week after chemo 2), and day 52-54 (10 days after chemo 4). (This might be subject to change in cases where the days of the chemo therapy are changed
  measuring the change in side effects side effects (expected) (31 questions): probability, intensity, coping, and compliance intention side effects (experienced)(21 questions): intensity, number, coping, compliance intention
psychological outcomes | Day 0 (day before chemo 1), day 7-10 (week after chemo 1), day 21-23 (week after chemo 2), and day 52-54 (10 days after chemo 4). (This might be subject to change in cases where the days of the chemo therapy are changed
  measuring the change in psychological outcomes communication satisfaction, trust, self-efficacy, distress (4 questions)
medical outcomes | day 54 (12 days after chemo 4). (This might be subject to change in cases where the days of the chemo therapy are changed
  use of co-medication (1 question)

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth van vliet, Principal Investigator — Leiden University
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
When giving consent participations are informed that i) for storage, analysis, publication, and archiving only coded research data will be used ii) and that the coded research data might be used for further or future analysis. Anonymized data might be shared on an Open Science platform.